CLINICAL TRIAL: NCT07400692
Title: Treatment of Olecranon Fractures in the Elderly, a Randomised Controlled Trial Comparing Surgical and Conservative Treatment
Brief Title: This is a Study to Find Out Whether Surgery Using a Metal Plate to Fix a Broken Elbow in Older Adults Leads to Better Recovery and Arm Function Compared to Non-surgical Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-049
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Olecranon Fracture
MeSH Terms: conditions — Olecranon Fracture | interventions — Open Fracture Reduction; Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery (Experimental): Open reduction and plate osteosynthesis. The surgical treatment will be performed with a direct approach to the olecranon using a locking compression plate.
  Interventions: Procedure: Open reduction and plate osteosynthesis
- rehabilitation (Other): Standard rehabilitation with optional upper arm sling for comfort for 2 weeks and progressive mobilization protocol
  Interventions: Other: Conservative treatment with early mobilisation

INTERVENTIONS:
Procedure: Open reduction and plate osteosynthesis — A cut is made along the back of the elbow to reach the broken bone. The surgeon carefully moves tissues aside and protects nearby nerves.
  The broken bone is cleaned, realigned, and held in place with a special metal plate and screws. This helps support the bone, especially in older patients with fragile bones. The surgeon checks the placement using live X-ray and moves the arm to ensure stability.
  The area is then closed with stitches, bandaged, and sometimes supported with a light splint. Recovery starts early, with gentle exercises to regain movement while protecting the repair.
  Arms: surgery
Other: Conservative treatment with early mobilisation — Conservativel treatment usually involves wearing a sling or light support for about two weeks to manage pain. After that, the patient begins gentle, supervised arm movements to prevent stiffness and muscle loss. As the pain improves, exercises become more active and focused on regaining strength. The goal is to let the bone heal while keeping the elbow working well.
  Arms: rehabilitation

SUMMARY:
This study takes place in one hospital and uses a random method to divide patients into groups. It looks at the best way to treat a broken elbow (specifically, a displaced olecranon fracture) in older adults who don't use their arms heavily. There are 84 patients in total, with 42 people in each group

ELIGIBILITY:
Inclusion Criteria

* Patients with an acute (< 2 weeks) Mayo type 2A or 2B olecranon fracture
* Patients aged > 65 years • Patients with reduced functional demand, with a score > 2 and < 7 on the Clinical Frailty Scale
* Patients able to provide informed consent and follow all study procedures as indicated in the protocol
* Signed informed consent for study participation

Exclusion criteria:

* Patients aged < 65 years or with a Clinical Frailty Scale score > 7 or < 2
* Patients with a Mayo type 2A or 2B fracture seen more than 2 weeks after injury
* Old fracture (> 6 months), pseudoarthrosis, or unhealed nerve injury of the ipsilateral upper limb
* Open (Gustilo-Anderson type 2 or 3) or pathological fracture
* Previous injury to, or other condition of, the elbow with severe functional impairment
* Patients with severe comorbidities preventing safe surgical treatment
* Other acute fracture or nerve damage of the ipsilateral upper limb
* Known drug or alcohol abuse
* Inability to follow study procedures (e.g., due to language barriers or severe comorbidities)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2030-02-03 (Estimated); Study Completion 2030-02-03 (Estimated)

PRIMARY OUTCOMES:
between-group difference in the Oxford Elbow Score (Italian Version) with the subscales Function, Pain, and Social-Psychological | 6 months after injury
  the Oxford Elbow Score is a patient-reported outcome measure specifically developed to evaluate elbow function. It includes 12 items divided into three domains: elbow pain, elbow function, and social-psychological impact. Each item is scored on a 5-point scale, and domain scores can be summed to obtain an overall score, where higher values indicate better outcomes. It is validated for use in both clinical and research settings and is sensitive to change, making it suitable for assessing treatment effects in patients with elbow disorders

CONTACTS AND LOCATIONS:
Overall Officials: Davide Previtali, MD, Principal Investigator — EOC
Locations (1):
- EOC - Orthopaedics and Traumatology Service, Lugano, Switzerland